CLINICAL TRIAL: NCT07394959
Title: Clinical Study on Tailored Hydration by Remote Dielectric Sensing System to Prevent Acute Renal Injury in Elderly Patients With Renal Insufficiency After Coronary Angiography
Brief Title: Hydration Guided by Remote Dielectric Sensing (ReDS) System for Preventing Acute Kidney Injury in Elderly Patients With Renal Insufficiency for Coronary Angiography and Intervention
Acronym: HISTORY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, MD, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ReDS guiding hydraton; 2024-17 (Other: Chinese PLA general hospital)
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Chronic Kidney Disease; Elderly
Keywords: contrast induced acute kidney injury; acute pulmonary edema
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored hydration guided by ReDS system (Experimental): The group guided by lung water monitor adjust hydration infusion rate dynamically adjusts based on the lung water parameters from the ReDS system.
  Interventions: Procedure: Tailored hydration guided by ReDS system
- Cntrol group (No Intervention): The control group performs the conventional hydration recommended by guidelines: administering normal saline at a rate of 1 ml/kg/h from 6 hours before procedure to 12 hours after procedure.

INTERVENTIONS:
Procedure: Tailored hydration guided by ReDS system — If initial lung water index is ≥35%, the hydration rate is 1ml/kg/h; If the initial lung water index is <35% but ≥20%, the hydration rate is 2ml/kg/h; If the initial lung water index is <20%, the hydration rate is designed to 5ml/kg/h. We re-check the lung water index after the contrast procedure. If the lung water index is >35% or if there is a more than 2-fold increase in the lung water index compared to pre-procedure, adjust the fluid infusion rate to 0.5ml/kg/h. If the lung water index after the contrast procedure is ≥20% but <35%, adjust the fluid infusion rate to 1ml/kg/h. If the lung water index after the contrast procedure is still <20%, adjust the fluid infusion rate to 5ml/kg/h.
  Arms: Tailored hydration guided by ReDS system

SUMMARY:
Explore the effectiveness and safety of tailored hydration guided by lung water index monitor system for prevention of acute kidney injury after percutaneous coronary intervention for elderly patients with renal insufficiency.

DETAILED DESCRIPTION:
The elderly patients with coronary heart disease is often complicated with chronic kidney disease, and these high risk patients has a risk of developing contrast induced acute kidney injury after undergoing percutaneous coronary intervention. Hydration is an important prevention to reduce the risk of contrast induced acute kidney injury , but hydration may cause acute left heart failure in elderly patients with renal insufficiency. We designed to give the elderly patients necessary hydration volume to reduce the risk of contrast induced acute kidney injury, and meanwhile avoid acute pulmonary edema caused by excessive preload. This study aimed to explore tailored hydration guided by lung water monitoring to prevent contrast induced acute kidney in elderly patients with renal insufficiency undergoing percutaneous coronary intervention. This study randomly divided elderly patients who are planning to undergo coronary intervention into two groups: tailored hydration group guided by remote dielectric sensing (ReDS system) and control group. The intervention group uses ReDS system to dynamically monitor the lung water index of enrolled patient, and fluid infusion rate is dynamically adjusted by lung water index to prevent the occurrence of acute pulmonary edema. We plan to evaluate the occurrence of postoperative acute kidney injury and acute pulmonary edema in two groups during the perioperative period. We follow up both major cardiovascular events and hemodialysis events in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;
* Patients with unstable angina pectoris are scheduled for percutaneous coronary intervention；
* Patients with chronic renal disease (estimated glomerular filtration rate < 90 ml/min);
* Sign the informed consent form.

Exclusion Criteria:

* 1. Acute decompensated severe heart failure or cardiogenic shock;
* 2. Malignant tumors, severe renal failure (estimated glomerular filtration rate < 30 ml/min);
* 3. Respiratory failure;
* 4. Used contrast media within one week;
* 5. Have allergic to contrast medium

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Contrast induced acute kidney injury | 3 days after procedure
  Increase in the creatinine level of at least 0.5 mg/dl (44 μmo/L) or at least a 25% increase from the baseline level within 2 to 3 days after PCI

SECONDARY OUTCOMES:
Acute kidney injury | 2 days after procedure
  An absolute increase in serum creatinine > 0.3mg/dl within 48 hours after percutaneous coronary intervention
Acute pulmonary edema | 7 days after procedure
  Dyspnea, significant increase in lung rales, accompanied by decreased oxygen saturation and significantly elevated brain natriuretic peptide
Renal replacement therapy | 12 months after procedure
  Hemodialysis or peritoneal dialysis
Persistent renal insufficiency | 3 months after procedure
  Glomerular filtration rate decreased by ≥25% compared to baseline 3 months after percutaneous coronary intervention
Cardiovascular adverse events | 12 months after procedure
  All-cause mortality, non-fatal acute myocardial infarction, unplaned revascularization for acute coronary syndrome ; readmission due to acute heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Mauler-Wittwer S, Sievert H, Ioppolo AM, Mahfoud F, Carrie D, Lipiecki J, Nickenig G, Fajadet J, Eckert S, Morice MC, Garot P. Study Evaluating the Use of RenalGuard to Protect Patients at High Risk of AKI. JACC Cardiovasc Interv. 2022 Aug 22;15(16):1639-1648. doi: 10.1016/j.jcin.2022.05.036. Epub 2022 Jul 27. PMID 35981838
- [Background] Maioli M, Toso A, Leoncini M, Micheletti C, Bellandi F. Effects of hydration in contrast-induced acute kidney injury after primary angioplasty: a randomized, controlled trial. Circ Cardiovasc Interv. 2011 Oct 1;4(5):456-62. doi: 10.1161/CIRCINTERVENTIONS.111.961391. Epub 2011 Oct 4. PMID 21972403
- [Background] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027
- [Background] Uriel N, Sayer G, Imamura T, Rodgers D, Kim G, Raikhelkar J, Sarswat N, Kalantari S, Chung B, Nguyen A, Burkhoff D, Abbo A. Relationship Between Noninvasive Assessment of Lung Fluid Volume and Invasively Measured Cardiac Hemodynamics. J Am Heart Assoc. 2018 Nov 20;7(22):e009175. doi: 10.1161/JAHA.118.009175. PMID 30571493
- [Background] Moroni F, Baldetti L, Kabali C, Briguori C, Maioli M, Toso A, Brilakis ES, Gurm HS, Bagur R, Azzalini L. Tailored Versus Standard Hydration to Prevent Acute Kidney Injury After Percutaneous Coronary Intervention: Network Meta-Analysis. J Am Heart Assoc. 2021 Jul 6;10(13):e021342. doi: 10.1161/JAHA.121.021342. Epub 2021 Jun 25. PMID 34169747
- [Background] Mohebi R, Karimi Galougahi K, Garcia JJ, Horst J, Ben-Yehuda O, Radhakrishnan J, Chertow GM, Jeremias A, Cohen DJ, Cohen DJ, Maehara A, Mintz GS, Chen S, Redfors B, Leon MB, Stuckey TD, Rinaldi MJ, Weisz G, Witzenbichler B, Kirtane AJ, Mehran R, Dangas GD, Stone GW, Ali ZA. Long-Term Clinical Impact of Contrast-Associated Acute Kidney Injury Following PCI: An ADAPT-DES Substudy. JACC Cardiovasc Interv. 2022 Apr 11;15(7):753-766. doi: 10.1016/j.jcin.2021.11.026. Epub 2022 Mar 16. PMID 35305904
- [Background] Feng W, Zhou J, Lun Z, Zhou D, Li P, Ye J. A Comparison Between Two Different Definitions of Contrast-Associated Acute Kidney Injury for Long-Term Mortality in Patients with Chronic Kidney Disease Undergoing Coronary Angiography. Clin Interv Aging. 2024 Feb 19;19:303-311. doi: 10.2147/CIA.S452882. eCollection 2024. PMID 38404478